CLINICAL TRIAL: NCT01835301
Title: Intra-stent Tissue Evaluation Within BMS and DES > 3 Years Since Implantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IntraStent
Record Dates: First submitted 2013-04-12; First posted 2013-04-18 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: In-stent Coronary Artery Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DES: Patients who received a DES stent > 3 years ago.
- BMS: Patients who received BMS stents > 3 years ago.

SUMMARY:
This study aims to test the hypothesis that plaque composition differs within a stent between bare metal stents and drug eluting stents (DES). It is possible that a difference in plaque composition seen within a stent may be contributory to the late thrombotic events seen more frequently with DES.

ELIGIBILITY:
Inclusion Criteria:

* Subject > 18 years of age;
* Subject, male or female, who underwent DES or BMS implantation in a native coronary vessel more than 3 year ago;
* Subject is scheduled for a diagnostic coronary or interventional procedure;
* Subject is willing to sign the informed consent.

Exclusion Criteria:

* Subject requires emergency catheterization;
* Subject has an acute myocardial infarction defined as anginal symptoms with ST-elevation on the EKG or creatine kinase-MB elevation >3times the upper limit of normal;
* Angiographic evidence of ≥ 70% stenosis within the target stent (visual estimate);
* Subject presented with cardiogenic shock;
* Subject has angiographically confirmed thrombus in the target coronary artery;
* Subject has a complex lesion not amenable to the IVUS/VH catheters and/or OCT catheters passing the stented segment;
* Subject has a contraindication to angiography/IVUS/OCT;
* Female subject is pregnant or lactating;
* Subject has life threatening comorbid conditions for which the investigator feels the subject should not be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 40 subjects will be enrolled in the study, with 20 patients who previously received BMS > 3 years ago and 20 patients who previously received DES > 3 years ago
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Plaque composition | During hospital stay, about 2 days.
  This study aims to test the hypothesis that plaque composition differs within the stent between BMS and DES. It is possible that a difference in plaque composition seen within the stent may be contributory to the late thrombotic events seen more frequently with DES.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Medstar Washington Hospital Center, Washington D.C., District of Columbia, United States